CLINICAL TRIAL: NCT06441682
Title: A Phase 2a, Double-Blinded, Randomized, Placebo-Controlled, and Active-Treatment Extension Study to Assess the Safety, Tolerability, Efficacy, Pharmacokinetics, and Immunogenicity of ARGX-119 in Participants With Amyotrophic Lateral Sclerosis
Brief Title: A Safety and Efficacy Study of ARGX-119 in Adult Patients With Amyotrophic Lateral Sclerosis (ALS)
Acronym: ReALiSe
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-119-2303; 2024-511318-19-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ARGX-119 - Dose 1 (Experimental): Participants will receive first dosage level of ARGX-119 intravenously during the double blinded treatment period followed by ARGX-119 in active treatment extension period
  Interventions: Biological: ARGX-119
- ARGX-119 - Dose 2 (Experimental): Participants will receive second dosage level of ARGX-119 intravenously during the double blinded treatment period followed by ARGX-119 in active treatment extension period
  Interventions: Biological: ARGX-119
- ARGX-119 - Dose 3 (Experimental): Participants will receive third dosage level of ARGX-119 intravenously during the double blinded treatment period followed by ARGX-119 in active treatment extension period
  Interventions: Biological: ARGX-119
- Placebo (Placebo Comparator): Participants will receive placebo intravenously during the double-blinded treatment period followed by ARGX-119 in active treatment extension period
  Interventions: Biological: ARGX-119; Other: Placebo

INTERVENTIONS:
Biological: ARGX-119 — Intravenous infusion of ARGX-119
Other: Placebo — Intravenous infusion of placebo
  Arms: Placebo

SUMMARY:
This study aims to evaluate the safety of ARGX-119 in adults with ALS. The study will also assess the impact of ARGX-119 on ALS disease outcomes, including muscle function. The study consists of 2 periods: a treatment period when participants will receive one of three ARGX-119 doses or placebo and an extension period when all participants will receive the same dose of ARGX-119. Participation in the study will last up to approximately 100 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participant is at least 18 and ≤80 years of age
* The participant is diagnosed with familial or sporadic ALS according to Gold Coast criteria
* The participant has a Treatment Research Initiative to Cure ALS (TRICALS) risk profile of ≥ -6.0 to < -2.0
* Slow vital capacity (SVC) of ≥ 60% of the predicted value according to Global Lung Function Initiative 2012

Exclusion Criteria:

* Use of noninvasive ventilation more than 10 hours a day or use of a tracheostomy for ventilatory support
* Any history of or current exposure to any gene or cell therapies (off-label use or investigational) for ALS
* Pregnant or lactating state or intention to become pregnant during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of adverse events (AEs) | Up to week 96

SECONDARY OUTCOMES:
Rate of change from baseline in electrophysiological muscle scan (MScan)-derived motor unit number (MUN) | Up to week 24
Maximum observed serum concentration (Cmax) of ARGX-119 | Up to week 96
Incidence of anti-drug antibodies (ADA) against ARGX-119 in serum over time | Up to week 96
Prevalence of anti-drug antibodies (ADA) against ARGX-119 in serum over time | Up to week 96

CONTACTS AND LOCATIONS:
Locations (9):
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - Kaye Edmonton Clinic, Edmonton
  - Montreal Neurological Institute and Hospital, Montreal
- Denmark (2):
  - Aarhus Universitets Hospital, Aarhus
  - Bispebjerg University Hospital, Copenhagen
- France (2):
  - Hôpital La Pitié Salpêtrière, Paris
  - CHU Bretonneau, Tours
- UMC Utrecht, Utrecht, Netherlands
- Akademiskt specialistcentrum Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No